CLINICAL TRIAL: NCT06244940
Title: The Sequencing for Detection in Congenital Heart Disease (SD-CHD) Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Scripps Translational Science Institute (Other)
Responsible Party: Principal Investigator, Rebecca Reimers, Principal Investigator, Scripps Translational Science Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-23-8202
Record Dates: First submitted 2023-10-28; First posted 2024-02-06 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Whole Genome Sequencing (WGC) from subject samples (Other)
  Interventions: Diagnostic Test: Whole Genome Sequencing (WGC) from subject samples

INTERVENTIONS:
Diagnostic Test: Whole Genome Sequencing (WGC) from subject samples — Perform whole genome sequencing (WGS) on fetuses with prenatally detected congenital heart disease (CHD) who meet inclusion criteria. Assess diagnostic yield of WGS in CHD and effect of prenatal versus postnatal phenotype on diagnostic yield.

SUMMARY:
This study is enrolling pregnant persons treated at Rady Children's Hospital fetal cardiology program with a prenatal diagnosis of congenital heart disease to look for genetic disorders in the fetus or unborn baby.

Congenital heart disease (CHD) is a group of structural differences to the heart that represent the most common birth defect among liveborn infants world-wide. CHD is the leading cause of birth-defect associated infant death. Prenatal detection allows for delivery planning, postnatal repair, specialized medications, and detailed counseling for parents. Up to one in three fetuses with CHD may have a genetic cause. In babies, knowing about genetic diseases helps patients and doctors provide the best care for their babies. If identified prenatally, this same knowledge may help participants prepare for their location of delivery, meet with specialists, and consider specialized treatments and medications that may be appropriate.

The diagnostic yield and clinical utility of whole genome sequencing (WGS) in fetuses with prenatally detected congenital heart disease (CHD) will be compared to routine clinical testing in patients choosing amniocentesis or chorionic villus sampling. DNA will be obtained from fetal samples and biological parent blood samples and analyzed according to standard clinical interpretation guidelines. Results will be reported to healthcare providers and patients and measures of clinical utility will be collected. Additionally, measures of stress, anxiety, depression, and perceived utility of information will be assessed by validated survey tools. A historical cohort of patients electing for diagnostic procedures will be used as a comparison population.

DETAILED DESCRIPTION:
Many genetic causes of CHD are missed by standard microarray and karyotype. Whole genome sequencing (WGS) and other specialized technologies for genetic and epigenetic diagnosis such as long-read sequencing, digital droplet PCR, RNA sequencing, and methylation analysis will identify additional causes of CHD but these technologies have not been systematically offered to patients prenatally.

Precision fetal diagnosis has expanded from diagnosis of aneuploidy on karyotype to copy number variants detected on microarray (such as 22q11 deletion syndrome) to gene sequencing through gene panels and exome sequencing (ES). Overall, prenatal ES in the setting of an ultrasound anomaly has had diagnostic yields of 8.5% and 10% in fetuses with normal microarray and karyotype. Anomaly-specific cohorts have noted diagnostic rates of up to 29% in nonimmune hydrops, an etiology with genetic heterogeneity and overlap with CHD. Uptake in ES in prenatal diagnosis has been limited by patient access due to cost, the time needed for testing, provider comfort with the broad nature of ES, and potential variants of uncertain significance and secondary findings.

The quality and accuracy of the data from genomic sequencing is directly related to quality and accuracy of information that goes into the bioinformatic analysis. One small study noted that when prenatal ES cases were reanalyzed postnatal or after autopsy results were available, an additional 20% of cases reached a diagnostic result due to the increased phenotypic information. The influence of phenotype on diagnostic yield of genomic sequencing for specific anomalies is unclear.

The importance of viewing the fetal and neonatal period as a continuum of care is increasingly recognized. Prenatal detection of critical CHD has the opportunity to help a family to optimize neonatal survival and learning of the other health challenges, or lack thereof, may have a large influence on parental preparedness. This may influence their levels of stress, and clinical management decisions such as what consultants to meet with prenatally, which center to choose for delivery, and potentially even what therapeutics to consider in the first months and years of life. A prior pediatric cohort of patients with hypertrophic cardiomyopathy (HCM) noted that among those with a new molecular diagnosis, 73% of individuals had a pathogenic variant identified in a gene with established clinical management recommendations, 36% were in syndromic HCM genes, and 2.9% were in genes with an eligible clinical trial.

Specific aims:

1. Perform whole genome sequencing (WGS) on fetuses with prenatally detected congenital heart disease (CHD) who meet inclusion criteria. Assess diagnostic yield of WGS in CHD and effect of prenatal versus postnatal phenotype on diagnostic yield.
2. Improve bioinformatic filtering and prenatal phenotyping for phenotype-causing gene identification through the use of detailed ultrasonographic examinations, magnetic resonance imaging, autopsy or pathology findings, and biochemical or proteomic profiling results when available.
3. Evaluate WGS utility on pregnancy and neonatal care including choice of delivery location, antenatal consultation with subspecialist providers, and postnatal interventions and consultation with subspecialist providers.

Through these aims, the study team will expand scientific understanding of genetic diagnosis in fetuses with CHD and will evaluate the impact on families anxiety, depression, and assess the clinical utility of this information. This information will allow for patient-centered approaches to implementing new technologies while improving the health outcomes and allowing for future disease-specific tailored care in the most common structural malformation identified on prenatal ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant individual with ongoing pregnancy with prenatally detected fetal CHD
* Desire for genetic diagnosis and clinical plan for amniocentesis or chorionic villus sampling

Exclusion Criteria:

* Gestational age of 38 weeks or greater
* Clinical course entirely explained by known chromosomal abnormality or confirmed genetic diagnosis that explains the clinical condition
* Pregnant persons under 18 years of age

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield of WGS in fetal congenital heart disease | Anticipated 200 trios in 2 years
  Trios with pathogenic or likely pathogenic sequencing results/ total number of trios.

SECONDARY OUTCOMES:
Diagnostic yield by type of CHD lesion | Anticipated 200 trios in 2 years
  As with primary outcome, diagnostic yield subcategorized into valvular defects, atrial and ventricular septal defects, inflow, and outflow tract anomalies
Patient utility of WGS as measured by: The Genome Empowerment Scale (GEmS) | Final survey 18 months after birth
  Used to measure the psychological impact and personal empowerment of receiving genomic test results in a wide range of clinical conditions. GEmS consists of 28 items and four derived factors. The four factors appear to assess the following dimensions: Factor 1 - Meaning of a diagnosis (parental perception of the utility of the genomic sequencing and importance of the resulting information); Factor 2 - Emotional management of the process (parental confidence in their ability to manage emotions related to the diagnostic process and outcome); Factor 3 - Seeking information and support (parental confidence in their ability to take the next steps to find new information and support); and Factor 4 - Implications and Planning (seeking health provider support and importance of information for family reproductive decisions). The higher the factor score, the stronger the participant is in each assessed dimension.
Patient utility of WGS as measured by: The Feelings About genomiC Testing Results (FACToR) Questionnaire | Final survey 18 months after birth
  Scored previously published, validated tools designed to be a brief, sensitive, and patient-centered. Used to measure the psychological impact and personal empowerment of receiving genomic test results in a wide range of clinical conditions. The instrument includes 12 items and 4 subscales (negative emotions, positive emotions, uncertainty, privacy concerns) with a 5-point Likert scale. 0=not at all, 1=a little, 2=somewhat, 3=a good deal, 4=a great deal.
Provider utility of WGS: Clinician-reported Genetic testing Utility InDEx (C-Guide) | Final survey 18 months after birth
  Scored, previously published metric to assess clinical utility of genetic testing in clinical practice. Of the 30 C-GUIDE items, 27 are scored from 0 to 2 and three are scored from -2 to 0 using item-specific fixed response options. An item score >0 indicates positive utility, an item scores <0 indicates negative utility ("disutility"), and item scores of 0 indicate no utility.
  Possible C-GUIDE total scores for each scoring strategy range from -2 to 32 for each PV, -4 to 48 for one PV plus one SV, and -6 to 54 for one PV plus one SV plus one PGx cluster. C-GUIDE is an ordinal scale and items are not weighted.
Patient depression and anxiety measures over time: GAD7 | Final survey 18 months after birth
  Measured by standardized instrument General Anxiety Disorder-7 (GAD7) Minimum score is 0; Maximum score is 21; the higher the score means worse, more anxiety
Patient depression and anxiety measures over time: EPDS | Final survey 18 months after birth
  Measured by standardized instrument Edinburgh Perinatal/ Postnatal Depression Scale (EPDS) Minimum score is 0; Maximum score is 30; the higher score means worse, more depression
Demographics of the cohort. | Duration of enrollment.
  Standardized metrics from the Clinical Sequencing Evidence-Generating Research (CSER) consortium.

CONTACTS AND LOCATIONS:
Locations (1):
- Rady Children's Institute for Genomic Medicine, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No